Official Title: A Phase 1, Open-Label, Positron Emission Tomography Study in Healthy Adult Subjects to Determine the Relationship Between Plasma Concentration and Brain Target Occupancy of ASN51 Following a Single Oral Dose

**NCT ID:** NCT06390098

Document Date: SAP Version 1.0: 17 November 2021

# **Statistical Analysis Plan**

Clinical trial protocol title: A Phase 1, Open-Label, Positron Emission Tomography Study in Healthy Adult Subjects to Determine the Relationship Between Plasma Concentration and Brain Target Occupancy of ASN51 Following a Single Oral Dose HMR code: 21-001 Sponsor code: ASN51-102 EudraCT no: 2021-001918-10 CRO details: **HMR** Cumberland Avenue London NW10 7EW Sponsor details: Asceneuron S.A. **EPFL Innobation Part** Bâtiment B, CH-1015 Lausanne, SWITZERLAND Issued: 17 November 2021 1 Version:

Protocol version 2.0, 19 May 2021

Based on:

Prepared by:

# **Table of Contents**

| | LIST OF ABBREVIATIONS4 | |
|---|---|---|
| | JATURES | |
| | RODUCTION | |
| STUI | OY OBJECTIVE(S) AND ENDPOINT(S) | |
| 4.1 | Study objective(s) | |
| | 4.1.1 Primary objective(s) | |
| | 4.1.2 Secondary objective(s) | |
| 4.2 | Study endpoint(s) | |
| | 4.2.1 Primary endpoint(s) | |
| | 4.2.2 Secondary endpoint(s) | |
| 4.3 | Statistical hypotheses | |
| | DY DESIGN | |
| TIMI | E AND EVENTS TABLE | 10 |
| PLA | NNED ANALYSES | 10 |
| 7.1 | Interim analyses | 10 |
| 7.2 | Final analysis | 10 |
| | 7.2.1 Persons responsible for analysis | 10 |
| SAM | PLE SIZE CONSIDERATIONS | 10 |
| 8.1 | Sample size assumptions | 10 |
| ANA | LYSIS POPULATIONS | 10 |
| 9.1 | Analysis datasets | 11 |
| DATA<br>11 | A DISPLAY TREATMENT AND OTHER SUBGROUP DESCR | RIPTORS |
| 10.1 | Conventions for summary statistics and data displays | 11 |
| DAT | A HANDLING CONVENTIONS | 12 |
| 11.1 | Premature withdrawal and missing data | 12 |
| 11.2 | Derived and transformed data | 12 |
| 11.3 | Assessment windows | 12 |
| 11.4 | Vital signs reference ranges | 13 |
| STUI | DY POPULATION | |
| 12.1 | Disposition of subjects | |
| 12.2 | Protocol deviations | |
| 12.3 | Demographic and baseline characteristics | |
| 12.3 | | |
| 12.4 | Treatment compliance | 14 |

| 13 | SAFE | ETY ANALYSES | .14 |
|---|---|---|---|
| | 13.1 | Extent of exposure | .14 |
| | 13.2 | Adverse events | .14 |
| | 13.3 | Deaths, serious adverse events and other significant adverse events | .15 |
| | 13.4 | Adverse events leading to withdrawal from the study | .15 |
| | 13.5 | Clinical laboratory evaluations | .15 |
| | 13.6 | Other safety measures | .15 |
| | | 13.6.1 Vital signs | 15 |
| | | 13.6.2 ECG | 15 |
| | | 13.6.3 Physical examination | 15 |
| | | 13.6.4 Columbia-Suicide Severity Rating Scale (C-SSRS) | 15 |
| 14 | PHA | RMACOKINETIC ANALYSES | .16 |
| | 14.1 | Pharmacokinetic concentration data | .16 |
| | 14.2 | Pharmacokinetic parameters | .16 |
| 15 | PHA | RMACODYNAMIC ANALYSES | .16 |
| | 15.1 | PET analysis data | .16 |
| 16 | REFI | ERENCES | .17 |
| 17 | ATT | ACHMENTS | .17 |
| | 17.1 | Table of contents for data display specifications | .17 |
| | 17.2 | Data display specifications | .22 |
| | | 17.2.1 Table outlines | 22 |
| | | 17.2.2 Figure outlines | 33 |
| | | 17.2.3 Listing outlines | 36 |
| APP | ENDIX | A: PHARMACOKINETIC ANALYSIS | .45 |
| 1 | CAL | CULATION METHODS | .45 |
| | 1.1 | Data handling conventions | .45 |
| | | 1.1.1 Missing and BLQ concentrations | 45 |
| | 1.2 | AUC calculations | .45 |
| | 1.3 | Lambda-z calculations | .45 |
| | 1.4 | Observed v predicted values | .46 |
| 2 | PAR | AMETER DEFINITIONS | .47 |
| | 2.1 | Plasma parameters | .47 |
| APP | ENDIX | B: SAMPLE PAGE LAYOUT | .49 |

#### 1 List of abbreviations

 $\lambda_z$ Terminal rate constant ΑE Adverse event **AUC** Area under concentration-time curve **AUC**<sub>inf</sub> AUC from time zero to infinity  $AUC_t$ AUC from time zero to time t **AUC**<sub>last</sub> AUC from time zero to last measurable concentration BMI Body mass index Below the limit of quantification **BQL** Confidence interval CI Maximum plasma concentration  $C_{max}$ **CRF** Case report form Clinical study report **CSR** Columbia-Suicide Severity Rating Scale C-SSRS Electrocardiogram **ECG** Heart rate HR **ICH** International Conference on Harmonization **IMP** Investigational medicinal product MedDRA Medical Dictionary for Regulatory Activities N Number of subjects Number of observations used in analysis n **PCI** Potential clinical importance PD Pharmacodynamic(s) Positron emission tomography **PET** Pharmacokinetic(s) PK Portion of the ECG from the beginning of the P wave to the beginning of PR the QRS complex, representing atrioventricular node function. Q1 Lower quartile Upper quartile Q3 The ORS complex of the ECG reflects the rapid depolarization of the right ORS and left ventricles. QT Portion of the ECG between the onset of the Q wave and the end of the T wave, representing the total time for ventricular depolarization and repolarization. QTc Corrected portion of the ECG between the onset of the Q wave and the end of the T wave, representing the total time for ventricular depolarization and repolarization. OTc interval with Bazett's correction method **OTcB** OTc interval with Fridericia's correction method **OTcF** RO Receptor occupancy Portion of the ECG between consecutive R waves, representing the RR ventricular rate SAD Single ascending dose Serious adverse event SAE SAP Statistical analysis plan Standard deviation SD Standard error of mean **SEM** Safety Review Committee SRC Terminal elimination half-life  $t_{\frac{1}{2}}$ 

 $\begin{array}{ll} TEAE & Treatment-emergent \ adverse \ event \\ t_{max} & Time \ to \ maximum \ plasma \ concentration \\ V_T & Regional \ total \ volume \ of \ distribution \end{array}$ 

WHO World Health Organisation

# 2 Signatures

The following persons have read and agreed the content of this Statistical Analysis Plan:



#### 3 Introduction

This statistical analysis plan (SAP) is based on the current trial protocol (version 2.0, 19 May 2021). Where statistical methods differ substantially between this SAP and the protocol, that will be identified in this document.

This SAP describes the datasets and the statistical methods to be used for the reporting and analysis of all data collected during the trial except the analysis of the PK-RO which will be done by Invicro.

If a future protocol amendment necessitates a substantial change to the statistical analysis of the trial data, this SAP will be amended accordingly. If, after database lock, additional analyses are required to supplement the planned analyses described in this SAP, those unplanned analyses will not be described in an amended SAP, but they will be identified in the integrated clinical study report (CSR). Any deviations from this SAP will be documented in the CSR.

This SAP has been written in consideration of the following guidelines:

- International Conference on Harmonization (ICH) E9, Guidance for Industry: Statistical Principles for Clinical Trials (ICH E9 1998)<sup>1</sup>; and
- ICH E3, Guidance for Industry: Structure and Content of Clinical Study Reports (ICH E3 1995)<sup>2</sup>.

Pharmacokinetic (PK) analysis will be done using WinNonlin v8.3 or higher on a Windows PC. Statistical analysis will be done using SAS <sup>®</sup> 9.4 or higher on a Windows PC.

# 4 Study objective(s) and endpoint(s)

# 4.1 Study objective(s)

## 4.1.1 Primary objective(s)

• To assess the brain O-GlcNAcase occupancy using [<sup>18</sup>F] IMA601 PET, following a single oral dose of ASN51

# 4.1.2 Secondary objective(s)

- To assess the relationship between the plasma concentration of ASN51, and the time-course of brain O-GlcNAcase occupancy using [18F]-IMA601 PET, following a single oral dose of ASN51
- To assess the single dose safety and tolerability of ASN51 in healthy adult subjects under fasted conditions

# 4.2 Study endpoint(s)

#### 4.2.1 Primary endpoint(s)

• Pharmacodynamic (PD): [<sup>18</sup>F]-IMA601 regional total volume of distribution (VT) at each brain scan.

## 4.2.2 Secondary endpoint(s)

- Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) up to follow-up
- Serious Adverse Events (SAEs) up to 4 weeks after last administration
- Laboratory tests
- Vital signs
- ECG
- Physical examination
- Pharmacokinetic (PK): plasma concentration of ASN51 at the time of each post-dose PET scan.
- PK/PD: relationship between ASN51 exposure and receptor occupancy.

# 4.3 Statistical hypotheses

The trial is an exploratory one, and there are no null hypotheses to be tested.

# 5 Study design

This is an open-label, adaptive-design PET study to investigate the occupancy of O-GlcNAcase by ASN51 after single oral doses in healthy adult male and female subjects (aged 25-55 years, inclusive). The study schema is depicted in Figure 2 of the protocol.

Up to 10 subjects will be enrolled. Each subject will have up to 3 imaging sessions, with one scan in each session. In the first imaging session, subjects will have 240 ml of water followed by a baseline PET scan approximately 2 h later. In the second and third imaging sessions, subjects will receive a single oral dose of ASN51 with 240 ml of water, followed by an ontreatment PET scan. Safety and pharmacokinetic data of the SAD study ASN51-101 will be assessed by the Safety Review Committee (SRC) prior to the dosing of the first subject(s) to determine the first dose level to be administered in session 2 after the baseline session 1 and the timing of the PET scans in relation to the study drug administration time. At most 2 subjects will be dosed on the same study day. For subsequent sessions, the dose level and the time of the PET scan in all imaging session 2 and 3 will be determined after review of the results from

the first on-treatment PET scan, including the PK data. Subjects will receive an intravenous dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan.

This study will have an adaptive design: to adequately evaluate the exposure versus receptor occupancy (RO) relationship, various doses of ASN51 of up to 85% of the highest well-tolerated dose level in the preceding SAD study ASN51-101, and the timing of on-treatment PET scans may be altered based on emerging data or study logistical requirements. On-treatment PET scans may be scheduled up to 48 h post-dose.

After each on-treatment PET scan, the SRC will review available RO, PK, safety and tolerability data, before selecting the dose and PET scan timings for imaging session 3. Arterial blood sampling will be done during each PET scan to quantify the parent tracer related radioactivity over the course of the PET scan, and to establish a tracer metabolite corrected plasma input function. The total arterial blood volume required for each tracer injection will not exceed 145 mL. Arterial cannulation and arterial blood sampling may be reduced or removed if analysis of PET data from previous subjects indicates that noninvasive analysis of the PET scan data can be done. If a non-invasive analysis is not possible, the use of an arterial cannula with each PET scan will continue through the study.

Subjects will be screened within 21 days before their baseline PET scan. Their on-treatment PET scans will be within 7 days of their baseline scan with an interval of 7–14 days between imaging sessions 2 and 3. Subjects will be confined for 72 h after the study drug administration in sessions 2 and 3. After the baseline scan in session 1 without study drug administration, subjects may leave the unit in the evening. In the case of a technical failure (such as unsuccessful tracer synthesis), subjects may be asked to attend an additional ontreatment imaging session, in which they will receive a third oral dose of ASN51. There will be at least 7 days between each dose of ASN51. Subjects will not have more than 3 PET scans or 3 doses of ASN51 during the study. Subjects will have a follow-up visit at the research unit 7 days (± 3 days) after imaging session 3 (Day 8).

#### 6 Time and events table

Please refer to Table 1 of the protocol, version 2.0, dated 19 May 2021

# 7 Planned analyses

# 7.1 Interim analyses

No interim analyses are planned.

# 7.2 Final analysis

The database will be locked once all subjects have completed the study, data have been entered, and queries resolved. The final analysis will be carried out following database lock.

## 7.2.1 Persons responsible for analysis

Statistician

# 8 Sample size considerations

# 8.1 Sample size assumptions

The trial is hypothesis generating, so no formal calculation of sample size is appropriate. The sample size of at most 10 subjects is considered adequate to allow modelling of the relationship between ASN51 plasma concentrations and the occupancy of O-GlcNAcase and is within the range generally accepted for PET studies. Enrolment of subjects into the study will be stopped as soon as the brain O-GlcNAcase occupancy versus ASN51 plasma concentrations is sufficiently characterized in opinion of the SRC.

# 9 Analysis populations

The following populations will be identified

All-treated set: This analysis set includes all randomised subjects who

received study drug (at least one dose).

Safety set: This analysis set includes subjects from the all-treated set who

had at least one safety assessment post-baseline. The safety set will be employed in the analysis of tolerability and safety

variables.

PET population: The PET population will consist of randomised subjects who

receive study medication, have a baseline PET scan, at least one post-baseline PET scan, and a PK result immediately

preceding PET scan.

PK analysis population:

The PK analysis population will consist of the subjects who provide evaluable data for the comparisons of interest. These subjects should have at least one quantifiable plasma concentration, should not have violated any major entry criterion likely to confound the PK analysis, and should not have deviated significantly from the protocol between enrolment and successful study completion.

In all populations, treatment will be assigned based upon the treatment subjects actually received.

The primary endpoint will be analysed using the PET population.

## 9.1 Analysis datasets

All analysis datasets will be based on observed data, except as outlined in Section 11.2.

# 10 Data display treatment and other subgroup descriptors

The treatment groups will be sorted in ascending dose order. When a total column is included, it immediately follows the treatment groups which it aggregates.

Listings of data will be sorted and displayed by treatment group, subject number, and also by date and time if applicable.

The treatment descriptions to be used on all tables and listings are:

| Treatment Groups |
|------------------|
| xx mg ASN51 |

# 10.1 Conventions for summary statistics and data displays

The minimum set of summary statistics for numeric variables will be: n, mean, standard deviation (or standard error mean [SEM]), median, minimum, and maximum. 95% confidence intervals (CI) will be presented where appropriate for data interpretation.

Categorical data will be summarised in frequency tables with n and percentage. Summaries of a categorical variable will include all recorded values.

The minimum and maximum values will be presented with the same number of decimal places as the raw data collected on the CRF (or to 3 significant figures for derived parameters less than 100 and as integers for values more than 99). The mean and percentiles (eg median, Q1, and Q3) will be presented using one additional decimal place. The standard deviation and standard error will be presented using two additional decimal places.

# 11 Data handling conventions

## 11.1 Premature withdrawal and missing data

All subjects who withdraw prematurely from the study or study drug will be included in the statistical analyses.

If a subject completes the treatment period but has missing data, then this will be made apparent in the subject listings. Missing data will not be imputed except for as outlined in Section 11.2.

If the study is prematurely discontinued, all available data will be listed and a review will be carried out to assess which statistical analyses are still considered appropriate.

Data collected at unscheduled time points during the study will not be used in the summaries or data analyses. They will be included in the listings.

If time information (ie hours and/or minutes) for adverse events (AEs) or concomitant medication is missing, but the day is present, then the time will be calculated in days. If date information is partial or missing, then any derived times (eg AE start time from last study medication) will be listed as missing.

Conventions for handling missing plasma concentrations are given in Appendix A: Pharmacokinetic Analysis.

#### 11.2 Derived and transformed data

Baseline will be considered to be the latest value obtained before study drug administration (eg Day 1, pre-dose; or Day –1 if not recorded at pre-dose; or screening if not recorded at pre-dose or on Day –1).

Laboratory data will be reported in standard units. Out-of-range laboratory tests may be repeated. If a test is out of-range at baseline and repeated before dosing, the latest repeat value before dosing will be used as baseline. However, if a test is out-of-range and repeated at any other time during the study, the out-of-range value (not the repeat value) will be included in statistical summaries.

Triplicate vital sign measurements will be made at screening and the mean of the three measurements for each subject will be used for analysis.

The PK parameters to be derived are given in Appendix A: Pharmacokinetic Analysis.

#### 11.3 Assessment windows

No assessment windows are defined for this report.

# 11.4 Vital signs reference ranges

The following vital signs ranges will be used:

| Vital Sign | Range |
|---------------------------------|-------------------|
| Seated systolic blood pressure | 90–140 mm Hg |
| Seated diastolic blood pressure | 50–95 mm Hg |
| Seated heart rate | 45–100 beats/min |
| Respiration rate | 10–16 breaths/min |
| Tympanic temperature | 35.5–37.8°C |

# 12 Study population

# 12.1 Disposition of subjects

The disposition of all subjects in the safety population will be summarised including: number of subjects randomised; number completing the study, by treatment; and number withdrawn from the study.

All subjects who withdraw or are withdrawn from the study will be listed, by treatment, with the reason for withdrawal.

A listing of analysis populations will be provided.

#### 12.2 Protocol deviations

Before closing the database, data listings will be reviewed to identify any significant deviations and determine whether the data should be excluded from any analysis populations.

Major protocol deviations include subjects who:

- Entered the study even though they did not satisfy the entry criteria.
- Met the criteria for withdrawal from the study but were not withdrawn.
- Received the wrong treatment or incorrect dose.
- Received an excluded concomitant therapy.
- Received investigational product(s) past the expiration date.

In addition, subjects with minor time deviations (measurements taken outside the allowable windows) will be identified. Allowable time windows for pharmacokinetic samples and other procedures are given in HMR Trial Procedures Summary.

## 12.3 Demographic and baseline characteristics

Demographic and baseline characteristics (eg physical examination, vital signs and ECGs) will be listed and summarised.

Subjects who take concomitant medication will be listed. All non-trial medication will be coded using the latest version of the World Health Organisation (WHO) Drug Global dictionary current at the time of the database lock (version September 2021 or higher).

Medical and surgical history will also be listed.

## 12.4 Treatment compliance

Dates and times of dosing will be listed.

# 13 Safety analyses

Summaries and listings of safety data will use the safety population.

# 13.1 Extent of exposure

The dates and times of treatment dosing will be listed to indicate exposure to the study medication.

#### 13.2 Adverse events

AEs will be coded using the version of the Medical Dictionary for Regulatory Activities (MedDRA) which is current at the time of database lock (version 24.0 or higher).

All AEs will be listed.

The number of subjects with at least one treatment-emergent adverse event (TEAE) per treatment will be tabulated by actual treatment and MedDRA system organ class. A TEAE is defined as an event emerging during treatment (having been absent pre-treatment) or that worsens after treatment<sup>1</sup>.

For each of the following, the number of TEAEs and the number of subjects with TEAEs will be summarised by treatment group:

- TEAEs, by system organ class and preferred term
- Drug-related ("related" as recorded by the investigator) TEAEs, by system organ class and preferred term

Subjects with more than one TEAE will be counted only once, at the greatest severity or causality, for each system organ class/preferred term. Multiple TEAEs in a subject will be counted once per system organ class and preferred term. AEs with missing severity and/or causality will be treated as severe and definitely related, respectively.

Summaries will be sorted by system organ class and decreasing total incidence of preferred term.

# 13.3 Deaths, serious adverse events and other significant adverse events

Deaths and serious adverse events (SAEs) will be listed separately (fatal events separate from non-fatal events). Other significant AEs, as identified by the investigator in the CRF, will be listed separately.

# 13.4 Adverse events leading to withdrawal from the study

AEs leading to withdrawal will be listed separately.

## 13.5 Clinical laboratory evaluations

Data from haematology, coagulation, urinalysis and clinical chemistry will be summarised by treatment.

Data from haematology, coagulation and clinical chemistry outside the normal range will be listed separately and summarised.

# 13.6 Other safety measures

#### 13.6.1 Vital signs

Vital signs evaluation at each planned assessment will be summarised by actual treatment.

Vital signs data outside of the normal range will be listed and summarised.

A separate listing of vital sign findings, classified as clinically significant by the investigator will also be provided.

#### 13.6.2 ECG

QT interval data will be presented using Fridericia's (QTcF) and Bazett (QTcB) corrections.

ECG variables will be summarised by treatment and time point.

QTcF and QTcB values > 450 msec, PR interval shortening < 120 msec, and PR interval prolongation >220 msec will be listed by treatment and timepoint and summarised. A separate listing of ECG findings classified as abnormal by the investigator will also be provided.

#### 13.6.3 Physical examination

Abnormal physical examination findings will be listed.

## 13.6.4 Columbia-Suicide Severity Rating Scale (C-SSRS)

Positive C-SSRS data will be listed.

# 14 Pharmacokinetic analyses

The PK parameters to be derived are given in Appendix : Pharmacokinetic analysis.

PK concentration data and PK parameter data will be summarised using the PK analysis population.

#### 14.1 Pharmacokinetic concentration data

The plasma concentrations and dose-normalised plasma concentrations of ASN51 will be listed and summarised by treatment.

Using actual sample times, linear and semi-logarithmic plasma concentration-time plots will be prepared by treatment and synoptic linear and semi-logarithmic dose-normalised plasma concentration-time plots of ASN51 will be prepared. Both Session 2 and Session 3 profiles will be included on the same plot. The same linear and logarithmic scales will be used for each subject. The linear and semi-logarithmic plots for a given subject will be presented on the same page.

Mean plasma concentration versus time plots will be presented for ASN51 per treatment (synoptic plot) (normal scale and log-linear scale).

Mean dose normalised plasma concentration versus time plots will be presented for ASN51 per treatment (synoptic plot) (normal scale and log-linear scale).

# 14.2 Pharmacokinetic parameters

The pharmacokinetic parameters of ASN51 will be listed and summarised by treatment.

If there is a quantifiable plasma concentration of the baseline PK sample of session 3, that value will be used in addition for the calculation of the PK parameters for session 2.

# 15 Pharmacodynamic analyses

# 15.1 PET analysis data

Start and end date of each PET scan will be listed together with the scan start/stop time and the Dose drawn up, Dose administered, Residual 1, and Residual 2.

[18F]-IMA601 regional total volume of distribution (V<sub>T</sub>) at each brain scan will be listed for each session and for change from baseline.

The RO values will be listed for sessions 2 and 3, respectively, together with the plasma concentration of ASN51 at the time of the start of each post-dose PET scan; which will be calculated by log-linear interpolation from the two closest PK data points by subject and treatment.

These concentration data will be transferred to Invicro for the PK-RO analysis. The PK-RO analysis will be provided by Invicro and sent to HMR for the inclusion in the CSR.

#### 16 References

- 1. International Conference on Harmonization, 1998. Statistical Principles for Clinical Trials ICH Harmonised Tripartite Guideline. Guidance for Industry, E9, FDA federal register, Vol 63, 1998, p49583. Available at: http://www.fda.gov/cder/guidance.
- 2. International Conference on Harmonization, 1995. Structure and Content of Clinical Study Reports ICH Harmonised Tripartite Guideline. Guidance for Industry, E3, FDA federal register, Vol 61, 1996, p37320. Available at: http://www.fda.gov/cder/guidance.
- 3. International Conference on Harmonisation, 2005. Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs. Concept paper, Guidance for Industry, E14, Center for Drug Evaluation and Research (CDER). Available at: http://www.fda.gov/cder/guidance/6922fnl.htm.
- 4. Julious, SA & Debarnot, CAM (2000) "Why are Pharmacokinetic Data Summarised by Arithmetic Means?", Journal of Biopharmaceutical Statistics, 10 (1), p55-71

#### 17 ATTACHMENTS

#### 17.1 Table of contents for data display specifications

For overall page layout refer to Appendix B: Sample page.

The numbering in the tables below will take precedence over the numbering in the shells.

The following tables and figures will be produced (templates provided in Section 17.2.1 and 17.2.2):

| Table | Description | Population | Source<br>Listing | Template<br>(Shells below) |
|---|---|---|---|---|
| 10.1 | Summary of subject disposition | Safety | 16.2.1.2<br>16.2.3.1 | T_SD1 |
| 14.1 | DEMOGRAPHIC DATA | | | |
| 14.1 | Summary of demographic characteristics | Safety | 16.2.4.1 | T DM1 |
| 14.2 | PHARMACOKINETIC DATA | | | |
| 14.2.1 | Summary of derived ASN51 plasma pharmacokinetic concentration-<br>time data (units) by treatment | PK Analysis | 16.2.6.1.1 | <u>T_PK1</u> |
| 14.2.2 | Summary of derived ASN51 plasma pharmacokinetic parameters by treatment | PK Analysis | 16.2.6.1.2 | <u>T_PK3</u> |
| 14.2.3 | Summary of log-transformed derived ASN51 plasma pharmacokinetic parameters by treatment | PK Analysis | 16.2.6.1.2 | <u>T_PK4</u> |
| 14.3 | SAFETY DATA | | | |
| 14.3.1.1 | Summary of treatment-emergent adverse events | Safety | 16.2.7.1 | T AE1 |
| 14.3.1.2 | Summary of drug-related treatment-emergent adverse events | Safety | 16.2.7.1 | <u>T_AE1</u> |
| 14.3.2.1 | Listing of fatal adverse events | Safety | 16.2.7.1 | L AE1 PG |
| 14.3.2.2 | Listing of non-fatal serious adverse events | Safety | 16.2.7.1 | L AE1 PG |
| 14.3.2.3 | Listing of other significant adverse events | Safety | 16.2.7.1 | L AE1 PG |
| 14.3.3 | Narratives of deaths, other serious and significant adverse events | Safety | | - |
| 14.3.4.1 | Summary of laboratory values outside the normal range by treatment | Safety | 16.2.8.1 | <u>T_LB1</u> |
| | and planned relative time | | 16.2.8.2 | |
| | | | 16.2.8.3 | |
| 14.3.4.2 | Summary of laboratory values outside the normal range by treatment | Safety | 16.2.8.1 | <u>T_LB3</u> |
| | | | 16.2.8.2 | |
| | | | 16.2.8.3 | |
| 14.3.5.1 | Summary of chemistry laboratory values | Safety | 16.4 | <u>T LB2</u> |
| 14.3.5.2 | Summary of haematology laboratory values | Safety | 16.4 | <u>T_LB2</u> |
| 14.3.5.3 | Summary of coagulation laboratory values | Safety | 16.4 | <u>T_LB2</u> |
| 14.3.5.4 | Summary of urinalysis results | Safety | 16.4 | <u>T UR1</u> |

| Table | Description | Population | Source<br>Listing | Template<br>(Shells below) |
|---|---|---|---|---|
| 14.3.6.1 | Summary of vital signs | Safety | 16.4 | <u>T_VS1</u> |
| 14.3.6.2 | Summary of vital signs outside the normal range by treatment, planned relative time and parameter | Safety | 16.2.9.1 | T VS2 |
| 14.3.7.1 | Summary of ECG values | Safety | 16.4 | T_EG2 |
| 14.3.7.2 | Summary of QTcF, QTcB and PR interval values outside the normal range by treatment, planned relative time and category | Safety | 16.2.9.3 | T EG3 |

| Figure | Description | Population | Source<br>Listing | Template<br>(Shells below) |
|---|---|---|---|---|
| 14.2 | PHARMACOKINETIC DATA | | | |
| 14.2.1 | Individual ASN51 plasma concentration-time plots (linear and semi-log) | PK Analysis | 16.2.6.1.1 | <u>F_PK1</u> |
| 14.2.2 | Individual ASN51 dose-normalised plasma concentration-time plots (linear and semi-log) | PK Analysis | 16.2.6.1.1 | <u>F PK1</u> |
| 14.2.3 | Mean (+/- SD) ASN51 plasma concentration-time plots (linear and semi-log) | PK Analysis | 16.2.6.1.1 | <u>F_PK2</u> |
| 14.2.4 | Mean (+/- SD) ASN51 dose-normalised plasma concentration-time plots (linear and semi-log) | PK Analysis | 16.2.6.1.1 | <u>F_PK2</u> |

The following abbreviated listings will be produced (templates provided in Section 17.2.3):

| Listing | Description | Template (Shells<br>below) |
|---|---|---|
| 16.2.1 | Study dates & disposition of subjects | |
| 16.2.1.1 | Listing of study dates | L SD1 PG |
| 16.2.1.2 | Listing of reasons for withdrawal | L SD2 PG |
| 16.2.2 | Protocol deviations | |
| 16.2.2.1 | Listing of subjects with inclusion/exclusion criteria deviations | L DV1 PG |
| 16.2.2.2 | Listing of subjects with time deviations | L TD1 PG |
| 16.2.2.3 | Listing of subjects with other protocol deviations | L DV2 PG |

| Listing | Description | Template (Shells below) |
|---|---|---|
| 16.2.3 | Analysis sets, including subjects excluded from analysis | below) |
| 16.2.3.1 | Listing of analysis populations | L AN1 PG |
| 16.2.4 | Demographic data & concomitant medication | |
| 16.2.4.1 | Listing of demographic characteristics | L DM1 PG |
| 16.2.4.2 | Listing of concomitant medications | L CM1 PG |
| 16.2.4.3 | Listing of medical and surgical history | L MH1 PG |
| 16.2.5 | Study drug administration | |
| 16.2.5.1 | Listing of exposure data | L EX1 PG |
| 16.2.6 | Pharmacokinetic and pharmacodynamics data | |
| 16.2.6.1.1 | Listing of ASN51 plasma pharmacokinetic concentration-time data | L PK1 PG |
| 16.2.6.1.2 | Listing of derived ASN51 plasma pharmacokinetic parameters | L PK4 PG |
| 16.2.6.1.3 | Individual ASN51 plasma concentration-time plots for estimation of λz, | <u>F_PK10</u> |
| 160601 | with regression line | T. DD.1 |
| 16.2.6.2.1 | Listing of regional total volume of distribution of [18F]-IMA601 data | <u>L_PD1</u> |
| 16.2.6.2.2 | Listing of receptor occupancy and plasma concentration data of ASN51 | <u>L PD2</u> |
| 16.2.7 | Adverse events | |
| 16.2.7.1 | Listing of all adverse events | L AE1 PG |
| 16.2.7.2 | Listing of serious adverse events | L AE1 PG |
| 16.2.7.3 | Listing of adverse events leading to withdrawal from study | <u>L_AE1_PG</u> |
| 16.2.8 | Laboratory values | |
| 16.2.8.1 | Listing of clinical chemistry data outside the normal range | L LB1 PG |
| 16.2.8.2 | Listing of haematology data outside the normal range | L LB1 PG |
| 16.2.8.3 | Listing of coagulation data outside the normal range | <u>L LB1 PG</u> |
| 16.2.9 | Vital signs, ECG variables, physical findings and C-SSRS | |
| 16.2.9.1 | Listing of vital signs outside the normal range | L VS1 PG |
| 16.2.9.2 | Listing of clinically significant vital signs | L VS2 PG |
| 16.2.9.3 | Listing of QTcF, QTcB and PR interval values outside the normal range | L EG1 PG |
| 16.2.9.4 | Listing of abnormal ECG findings | L EG2 PG |
| 16.2.9.5 | Listing of abnormal physical examination findings | L PE1 PG |

| Listing | Description | Template (Shells |
|---|---|---|
| | | below) |
| 16.2.9.6 | Listing of positive Columbia-Suicide Severity Rating Scale data | L CSS PG |

Complete listings of all data collected in this study will also be produced.

# 17.2 Data display specifications

## 17.2.1 Table outlines

Note: Summary statistics for continuous data will only be provided for treatments where n>1

#### Template T\_SD1

Table 10.1 Summary of subject disposition

| | | | Treatment 1 | Treatment 2 | | All Subjects |
|---|---|---|---|---|---|---|
| Population | Status | Reason for Withdrawal | (N=xx) | (N=xx) | Etc | (N=xx) |
| | | | n (%) | n (%) | | n (%) |
| All-treated | Included | | xx (xx) | xx (xx) | | xx (xx) |
| Safety | Included | | XX | XX | | XX |
| | Completed | | xx (xx) | xx (xx) | | xx (xx) |
| | Withdrawn | | | | | |
| | | Death | xx (xx) | xx (xx) | | xx (xx) |
| | | Adverse Events | xx (xx) | xx (xx) | | xx (xx) |
| | | Withdrawal by subject | xx (xx) | xx (xx) | | xx (xx) |
| | | Study terminated by | xx (xx) | xx (xx) | | xx (xx) |
| | | Sponsor | | | | |
| | | Lost to follow-up | xx (xx) | xx (xx) | | xx (xx) |
| | | Other | xx (xx) | xx (xx) | | xx (xx) |
| Alternative 1 (if applicable) | Included | | | | | |
| Alternative 2 (if applicable) | Included | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups

Remove column "Reason for Withdrawal" if no subject withdrew

Add a footnote about n=4 for the dose group

#### Template T\_DM1

Table 14.1 Summary of demographic characteristics

| Variable | Statistics | All Subjects (N=xx) |
|---------------|----------------------------|---------------------|
| Age (y) | n | |
| | Mean | |
| | SD | |
| | Median | |
| | Min | |
| | Max | |
| Sex (%) | Female | |
| | Male | |
| Race (%) | American Indian or Alaskan | |
| | Native | |
| | Asian | |
| | Black | |
| | Native Hawaiian or other | |
| | Pacific Islander | |
| | White | |
| | Other | |
| Ethnicity (%) | Hispanic or Latino | |
| | Not Hispanic or Latino | |
| Height (cm) | n | |
| | Mean | |
| | SD | |
| | Median | |
| | Min | |
| | Max | |
| Weight (kg) | n | |
| | Mean | |
| | SD | |
| | Median | |
| | Min | |
| | Max | |

| Variable | Statistics | All Subjects (N=xx) |
|--------------|------------|---------------------|
| BMI (kg/m2) | n | |
| | Mean | |
| | SD | |
| | Median | |
| | Min | |
| | Max | |
| Smoker | Former | |
| History (%) | Never | |
| Alcohol* | n | |
| (units/week) | Mean | |
| | SD | |
| | Median | |
| | Min | |
| | Max | |
| Caffeine* | n | |
| (cups daily) | Mean | |
| | SD | |
| | Median | |
| | Min | |
| | Max | |
| Optional | | |
| (units) | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups and additional demographic characteristics

<sup>\*</sup>includes only those subjects who drink caffeine/alcohol

#### Template T\_PK1

Table 14..2.xx Summary of derived ASN51 plasma pharmacokinetic concentration-time data [units] by treatment

| Treatment | {Add.<br>time<br>var.} | Planned<br>Relative<br>Time | n | No.<br>Imputed | Mean | 95% CI<br>(Lower,Upper) | SD | %CVb | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | , | | | | | |
| Treatment 1 | | Pre-dose | Х | Х | XXXX.X | (xxxx.x,xxxx.x) | | XX.X | XXXX.X | XXXX | XXXX |
| (N=xx) | | 30 min | X | X | xxxx.x | (xxxx.x,xxxx.x) | XX.XX | XX.X | XXXX.X | XXXX | XXXX |
| | | 1 hr | x | X | XXXX.X | (xxxx.x,xxxx.x) | xx.xx | xx.x | XXXX.X | XXXX | xxxx |
| Treatment 2 | | Pre-dose | х | x | xxxx.x | (xxxx.x,xxxx.x) | xx.xx | XX.X | xxxx.x | xxxx | XXXX |
| (N=xx) | | 30 min | x | x | XXXX.X | (xxxx.x,xxxx.x) | xx.xx | xx.x | xxxx.x | xxxx | xxxx |
| | | 1 hr | х | X | xxxx.x | (xxxx.x,xxxx.x) | XX.XX | XX.X | xxxx.x | xxxx | XXXX |

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels and timepoints

#### Template T\_PK3

Table 14..2.xx Summary of derived ASN51 plasma pharmacokinetic parameters by treatment

| | | {Additional | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | time | | | 95% CI | | | | | |
| Parameter | Treatment | variables} | n | Mean | (Lower,Upper) | SD | %CVb | Median | Min | Max |
| AUC <sub>t</sub> (units) | Treatment 1 (N=xx) | | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | XX.X | XXXX.XX | xxxx.x | xxxx.x |
| | Treatment 2 (N=xx) | | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | XX.X | XXXX.XX | xxxx.x | xxxx.x |
| C <sub>max</sub> (units) | Treatment 1 (N=xx) | | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | XX.X | XXXX.XX | xxxx.x | xxxx.x |
| | Treatment 2 (N=xx) | | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | xx.xxx | xx.x | XXXX.XX | xxxx.x | xxxx.x |

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels, timepoints and parameters

Template T\_PK4

Table 14..2.xx Summary of log-transformed derived ASN51 plasma pharmacokinetic parameters by treatment

| Parameter | Treatment | {Additional time variables} | n | Geom<br>Mean | 95% Cl<br>(Lower,Upper) | SD (logs) | %CVb |
|---|---|---|---|---|---|---|---|
| AUC <sub>last</sub> (units) | Treatment 1 (N=xx) | | | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | xx.xx |
| | Treatment 2 (N=xx) | | | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | xx.xx |
| C <sub>max</sub> (units) | Treatment 1 (N=xx) | | | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | xx.xx |
| | Treatment 2 (N=xx) | | | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | xx.xx |

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels, timepoints and parameters

#### Template T\_AE1

Table 14.3.3.xx Summary of treatment-emergent adverse events

| | | Treatment 1 (N=xx) | Treatment 2 (N=xx) | Etc | All Subjects<br>(N=xx) |
|---|---|---|---|---|---|
| System Organ Class | Preferred Term | n (%) | n (%) | | |
| Number of subjects with TEAEs | | x (xx.x) | x (xx.x) | | |
| Gastrointestinal disorders | Total number of subjects | x (xx.x) | x (xx.x) | | |
| | Abdominal discomfort | x (xx.x) [xx] | x (xx.x) [xx] | | |
| | Abdominal pain $\downarrow$ | x (xx.x) [xx] | x (xx.x) [xx] | | |
| Nervous system disorders | Total number of subjects | | | | |
| | Dizziness | | | | |
| | Headache | | | | |
| | $\downarrow$ | | | | |
| $\downarrow$ | $\downarrow$ | | | | |

Source: Listing 16.2.xx

n = number of subjects (subjects with >1 TEAE are counted only once per system organ class and preferred term)

[] = number of TEAEs

Coded using MedDRA v xx.x

Programming notes: Continued with all treatment groups

SOCs and PTs are sorted in decreasing order of frequency

Presented for all applicable MedDRA system organ classes and terms.

#### Template T\_LB1

Table 14.3.4.xx Summary of laboratory values outside the normal range by treatment, planned relative time

| | | Planned Relative |
|---------------------|-----------|------------------|
| ratory Test (units) | Treatment | Time |

Laboratory Test (units)

Treatment 1 (N=xx)

Time m H L

Source: Listing 16.2.xx

H = Above reference interval, L = Below reference interval m = number of subjects with results for that parameter

*Programming notes:* Continued with all tests, treatment groups and time points.

#### Template T\_LB3

Table 14.3.4.xx Summary of laboratory values outside the normal range by treatment

| Laboratory Test (units) | Treatment | m | Н | L | Overall* |
|-------------------------|--------------------|---|---|---|----------|
| | Treatment 1 (N=xx) | | | | |

Source: Listing 16.2.xx

H = Above reference interval, L = Below reference interval Subjects only counted once per treatment per double flag

\*Subjects only counted once per treatment

*m* = total number of results for that parameter

*Programming notes:* Continued with all tests, treatment groups and time points.

#### Template T\_LB2

Table 14.3.5.xx Summary of chemistry laboratory values

| | | | | | | | | | | Ch | ange f | rom Baselin | ie | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Test | | Planned | | | | | | | | | | | | |
| (units) | Treatment | <b>Relative Time</b> | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| | Treatment 1 (N=xx) | | | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatments and time points

#### Template T\_UR1

Table 14.3.5.xx Summary of urinalysis results

| | Planned Relativ | e | Treatment | 1 (N=xx) | Treatment 2 (N=xx) | |
|---|---|---|---|---|---|---|
| Laboratory Test | Time | Result | n | (%) | n | (%) |
| | Time 1 | Positive | Х | Х | | |
| | | Negative | Х | Χ | | |
| | | Not Done | x | | | |
| | Time 2 | Positive | | | | |
| | | Negative | | | | |
| | | Not Done | | | | |

Source: Listing 16.2.xx

Programming notes: Results recorded as received, e.g. Negative, Trace, etc; urine pH summarised as <5, 5-8, >8; specific gravity summarised as <=1.005, 1.006-1.010, 1.011-1.015, 1.016-1.020, 1.021-1.025, 1.026-1.029, >=1.030 Continued with all treatment groups and time points

#### Template T\_VS1

Table 14.3.6.xx Summary of vital signs

| | | Planned | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable (units) | Treatment | Relative Time | n | Mean | SD | Median | Min | Max |
| Systolic BP (mmHg) | Treatment 1 (N=xx) | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all variables, treatments and time points

#### Template T\_VS2

Table 14.3.6.xx Summary of vital signs outside the normal range by treatment, planned relative time and parameter

| | Planned Relative | Systolic<br>Pressure | | | ic Blood<br>e (mmHg) | | t Rate<br>s/min) | Temper | ature (C) | e | tc |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Time | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| Treatment 1 | Time 1 | | | | | | | | | | |
| (N=xx) | Time 2 | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatments and parameters. n = total number of results for that parameter

#### Template T\_EG2

Table 14.3.7.xx Summary of ECG values

| | | Planned Relative | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable (units) | Treatment | Time | n | Mean | SD | Median | Min | Max |
| Heart Rate (bpm) | Treatment 1 (N=xx) | | | | | | | |
| | Treatment 2 (N=xx) | | | | | | | |
| PR Interval (msec) | Treatment 1 (N=xx) | | | | | | | |
| | Treatment 2 (N=xx) | | | | | | | |
| | | | _ | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups and time points

Do not summarise RR or QRS axis

#### Template T\_EG3

Table 14.3.7.xx Summary of QTcF, QTcB and PR interval values outside the normal range by treatment, planned relative time and category

| | | | QTcF (msec) | | | | | QTcB (msec) | | | | | PR int. (msec) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned<br>Relative | 451 | <b>-</b> 480 | 481 – 500 | | > 500 | | 451 – 480 | | 481 – 500 | | > 500 | | <120 | | >220 | |
| Treatment | Time | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| Treatment 1 | Time 1 | | | | | | | | | | | | | | | | |
| (N=xx) | Time 2 | | | | | | | | | | | | | | | | |
| | Time 3 | _ | | | | | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all variables, treatments and time points. n = total number of results for that parameter

# 17.2.2 Figure outlines

#### Template F\_PK1

Figure 14.2.xx Individual ASN51 plasma concentration-time plots (linear and semi-log)





Source: Listing 16.2.xx

Programming notes: For dose-normalised plot, the y-axis label will be "Dose-normalised concentration (units)"

#### Template F\_PK2

Figure 14.2.xx Mean (+/- SD) ASN51 plasma concentration-time plots (linear and semi-log)



Source: Listing 16.2.xx

BLQ values are imputed to zero

Programming notes: Offset treatment groups (to both sides of timepoint) to minimise overlapping error bars

#### Template F\_PK10

Figure 16.2.xx Individual ASN51 plasma concentration-time plots for estimation of lambda-z, with regression line



Source: Listing 16.2.xx
### **17.2.3** Listing outlines

#### Template L\_SD1\_PG

Listing 16.2.x.xx Listing of study dates

Subject Sequence\* Screening Period 1 Period 2 Period 3 Follow Up

Programming notes: Lists dates for screening, each dosing period and follow up

Add footnotes for the sequences

#### Template L\_SD2\_PG

Listing 16.2.x.xx Listing of reasons for withdrawal

Date of Study
Treatment Subject Withdrawal Day Reason

Programming notes: Reason for withdrawal is concatenation of reason and details

#### Template L\_DV1\_PG

Listing 16.2.x.xx Listing of subjects with inclusion/exclusion criteria deviations

Treatment Subject Type Criterion

Inclusion
Exclusion

Sponsor code: ASN51-102

#### Template L\_TD1\_PG

Listing 16.2.x.xx Listing of subjects with time deviations

| | | Planned | | Allowed | Actual | Time outside the |
|---|---|---|---|---|---|---|
| | | Relative | | deviation | deviation | deviation window |
| Treatment | Subject | Time | Procedure | (h:min) | (h:min) | (h:min) |

Programming notes: Only include time deviations which exceed the allowed deviation

#### Template L\_DV2\_PG

Listing 16.2.x.xx Listing of subjects with other protocol deviations

<u>Treatment</u> <u>Subject</u> <u>Protocol Deviation</u> <u>Type of Deviation</u> <u>Category</u>

#### Template L\_AN1\_PG

Listing 16.2.x.xx Listing of analysis populations

Safety

<u>Treatment Subject Population Population 1 Population 2 Etc.</u>

#### Template L\_DM1\_PG

Listing 16.2.x.xx Listing of demographic characteristics

| | | | | Age | | | | Height | Weight | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Sequence* | Date of visit | Year of birth | (y) | Sex | Race | Ethnic origin | (cm) | (kg) | BMI (kg/m2) Etc (units) |

\*A = 0 mg ASN51, B = xx mg ASN51, C = xx mg ASN51, D = xx mg ASN51,

Programming notes: A by-subject listing of demographic characteristics including:

Treatment

Subject

Date of visit

Year of birth

Age

Sex

Race / Ethnic Origin

Height (if collected only once during the study)

Weight (if collected only once during the study)

Smoking History

Alcohol Consumption

Additional study-specific demography characteristics included on the CRF

#### Template L\_CM1\_PG

Listing 16.2.x.xx Listing of concomitant medications

Study Day

Started/

ATC Class/ Drug Name/ Ongoing Dose/ Date/Time Started/ Time Since Last Started Pre-Medication Code\* Indication Freq/Route **Date Stopped** Trial? Medication? Treatment Subject Dose

Programming notes: \* only include this column and the footnote if coding used

Subject

Category

Include dose and units (e.g.

#### Template L\_MH1\_PG

Listing 16.2.x.xx Listing of medical and surgical history

Treatment

System organ

class\*/Preferred Clinical Date Date End relative term Verbatim text significance Started Stopped to Screening

#### Template L\_EX1\_PG

Listing 16.2.x.xx Listing of exposure data

Start Date/ Dose Formulation/
Treatment 1 Subject Start Time of Dose Unit Route Frequency

Zanday

<sup>\*</sup>Coded using WHODrug Global vXX.X

<sup>\*</sup>Coded using MedDRA vXX.X

#### Template L\_PK1\_PG

Listing 16.2.6.xx Listing of ASN51 plasma pharmacokinetic concentration-time data

| | | {Add. | | | | | | Actual Relative | |
|---|---|---|---|---|---|---|---|---|---|
| | | time | | | Planned | Actual time | Time Deviation | Time | |
| Treatment | Subject | var.} | Date | Study Day | <b>Relative Time</b> | (hh:mm) | (min) | ( h) | Concentration (units) |

Below the Limit of Quantification (BLQ) is < xx units (e.g. 1 ng/mL)

Programming notes: Values below LLOQ are shown as BLQ. Check LLOQ value in final PK spreadsheet for each analyte.

#### Template L\_PK4\_PG

Listing 16.2.xx Listing of derived ASN51 plasma pharmacokinetic parameters

| | | Imaging | AUC <sub>inf</sub> | $AUC_t$ | $C_{max}$ | t <sub>1/2</sub> | $t_{max}$ |
|---|---|---|---|---|---|---|---|
| Treatment | Subject | Session | (units) | (units) | (units) | (units) | (units) |

Programming notes: Continue with all parameters

#### Template L\_PD1

Listing 16.2.xx Listing of [18F]-IMA601 data regional total volume of distribution

| | | | {Add. | Start Date/ | Stop Date/ | Dose | | | | | Change from |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Scan | time | Start Time of PET | Stop Time of | drawn | | | | $V_T$ | baseline V <sub>™</sub> |
| Treatment | Subject | number | var.} | scan | PET scan | up | Residual 1 | Residual 2 | Brain Region | (units) | (units) |

#### Template L\_PD2

Listing 16.2.xx Listing of receptor occupancy and plasma concentration data of ASN51



Programming notes: Concentration at start of PET scan will be calculated using the closest time before start of PET scan and the closest time after PET scan

#### Template L\_AE1\_PG

Listing 16.2.x.xx Listing of all adverse events

| | | | Outcome/ | | | Frequency/ | Related to Study |
|---|---|---|---|---|---|---|---|
| | | System Organ Class* / | Onset Date/Time/ | Study Day Started/ | Severity/ | Action Taken (1)/ | Drug/ |
| | | Preferred Term/ | Resolved Date/Time/ | Time Since Last | Serious/ | Other Action | Treatment |
| Treatment | Subject | Verbatim Text | Duration | Dose | Withdrawal | Taken | Emergent? |
| Treatment 1 | | Gastrointestinal Disorders / | Resolved/ | Day x/ | Mild/ | Intermittent/ Dose | Possibly/ |
| | | Intestinal Spasm / | | 10d 7h 3m | No/ | not changed/ | Yes |
| | | Entero-spasm | | | Yes | None | |
| | | | 34d 4h 5m | | | | |

(1) Action Taken with Study Treatment \*Coded using MedDRA vXX.X

Programming notes: For the listing of "other significant AES" include (from ICH E3) AEs leading to withdrawal, AEs leading to dose reduction (including drug withdrawn, interrupted, reduced or similar) and AEs with AEOSE=Y. If AEOSE has not been collected then use "Otherwise significant" in the CRF.

#### Template L\_LB1\_PG

Listing 16.2.x.xx Listing of clinical chemistry data outside the normal range

| | | | Planned<br>Relative | | Study | | | | Clinically |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Laboratory test (units) | Time | Date/Time | Day | Value | Reference Interval | RI | Significant? |
| Treatment 1 | | Alk Phos (U/L) | Time 1 | | -1 | 64.00 | 32.0 - 92.0 | | |
| | | | Time 2 | | 85 | 84.00 | 32.0 - 92.0 | | |
| | | ALT (U/L) | Time 1 | | -1 | 29.00 | 10.0 - 40.0 | | |
| | | | Time 2 | | 85 | 70.00 | 10.0- 40.0 | Н | Υ |

RI for Reference Interval flag;

H = Above reference interval, L = Below reference interval

Programming notes: Lists only subjects with at least a high or low value

#### Template L\_VS1\_PG

Listing 16.2.x.xx Listing of vital signs outside the normal range

| | | | | Systolic | Diastolic | |
|---|---|---|---|---|---|---|
| | | Planned Relative | | <b>Blood Pressure</b> | Blood Pressure | Etc |
| Treatment | Subject | Time | Date/Time | (mmHg) | (mmHg) | (units) |
| | | 24 H | | 63 | 148* | |

<sup>\*</sup> Value outside the normal range

#### Template L\_VS2\_PG

Listing 16.2.x.xx Listing of clinically significant vital signs

| | | Planned Relative | | | Comment on Clinical |
|---|---|---|---|---|---|
| Treatment | Subject | Time | Date/Time | Vital Sign Finding | Significance |

Programming notes: Lists only values with abnormal CS

#### Template L\_EG1\_PG

Listing 16.2.x.xx Listing of QTcF, QTcB and PR interval values outside the normal range

| | | 24 H | | 63 | 148 | 78 | 50 | 390 | 452* | 396 |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Relative Time | Date/Time | (bpm) | (msec) | (msec) | (deg) | (msec) | (msec) | (msec) |
| | | Planned | | Rate | PR Int. | Dur. | Axis | QT Int. | QTcF | QTcB |
| | | | | Heart | | QRS | QRS | | | |

<sup>\*</sup> Value outside the normal range

#### Template L\_EG2\_PG

Listing 16.2.x.xx Listing of abnormal ECG findings

| | | Planned Relative | | Comment on Clinical | |
|---|---|---|---|---|---|
| Treatment | Subject | Time | Date | ECG Finding | Significance |

Programming notes: Lists only values with Normal variant='No' or with comment on ECG result

ECG Finding contains Physician's Opinion from CRF and relates to whole trace (not individual parameters), e.g. Normal, Abnormal - NCS or Abnormal - CS

#### Template L\_PE1\_PG

Listing 16.2.x.xx Listing of abnormal physical examination findings

Planned Relative

Treatment Subject Time Date Site Details

Programming Notes: List only findings with an 'abnormal' result.

If subjects have multiple abnormal sites at a given time, create a separate row for each site.

#### Template L\_CSS\_PG

Listing 16.2.x.xx Listing of positive Columbia-Suicide Severity Rating Scale data

Planned Relative

Treatment Subject Time Date/Time Category Question Result

## Appendix A: Pharmacokinetic analysis

#### 1 Calculation methods

## 1.1 Data handling conventions

#### 1.1.1 Missing and BLQ concentrations

No missing values will be imputed.

For all PK assessments (calculation of parameters, and individual profile plots) BQL values will be taken as missing with the exception of the predose value, where a BLQ value will be taken as zero.

BQL values will be taken as zero for calculation of plasma concentration summary statistics unless they fall between two quantifiable concentrations in which case they will be treated as missing.

#### 1.2 AUC calculations

The AUC will be calculated by a combination of linear and logarithmic methods. The linear trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations.

It is acceptable to include data from profiles with >20% extrapolated as long as at least 80% of the profiles in the study have <20% of the  $AUC_{(0-\infty)}$  as extrapolated area. In this instance, individual plasma concentration-time profiles for which the extrapolated areas are >20% of  $AUC_{(0-\infty)}$  will be identified.

It is <u>unacceptable</u> to use  $AUC_{(0-\infty)}$  data if >40% of the AUC has been extrapolated, except in specific situations which should be carefully justified in the study report.

#### 1.3 Lambda-z calculations

The apparent terminal phase rate-constant  $(\lambda_z)$  will be estimated by linear regression of logarithmically transformed concentration versus time data. Only those data points

which are judged to describe the terminal log-linear decline will be used in the regression.

During the analysis, repeated regressions are carried out using the last three points with non-zero concentrations, then the last four points, last five, etc. Points prior to  $C_{max}$  are not used. Points with a value of zero for the concentration are excluded. For each regression, an adjusted  $R^2$  is computed. The  $\lambda_z$  using the regression with the largest adjusted  $R^2$  is selected. If the adjusted  $R^2$  does not improve, but is within 0.0001 of the largest adjusted  $R^2$  value, the regression with the larger number of points is used.  $\lambda_z$  must be positive, and calculated from at least three data points.

A minimum number of three data points will be used in calculating  $\lambda_z$ .

### 1.4 Observed v predicted values

For parameters dependent on  $\lambda_z$ , the 'predicted' rather than the 'observed' parameters will be calculated.

The 'predicted' parameters are calculated using  $\hat{C_t}$  (the predicted value of the concentration at time tn); whilst the 'observed' parameters use the last observed concentration.

## 2 Parameter definitions

# 2.1 Plasma parameters

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| Concentrations and | times | | | | | | |
| C <sub>max</sub> | Maximum (peak) plasma concentration | Obtained directly from the concentration-time data. | ng/mL | Y | Cmax | CMAX | C <sub>max</sub> |
| C <sub>max</sub> /Dose | Dose-normalised AUC to infinity | Calculated as C <sub>max</sub> /Dose administered | (ng/mL)/mg | Y | Cmax_D | CMAXD | C <sub>max</sub> /D |
| t <sub>max</sub> | Time to reach maximum (peak) plasma concentration | Obtained directly from the concentration-time data. | h | N | Tmax | TMAX | t <sub>max</sub> |
| Half-life | | | | | | | |
| $\lambda_z$ | Terminal rate constant | Estimated by linear regression of logarithmically transformed concentration versus time data. | 1/h | Y | Lambda_z | LAMZ | $\lambda_z$ |
| t <sub>½</sub> | Terminal half-life | Calculated from the terminal slope of the log concentration-time curve, as follows: $t_{1/2} = \frac{\log_e 2}{\lambda_z}$ | h | Y | HL_Lambda_z | LAMZHL | t <sub>1/2</sub> |
| Areas under the cur | ve | | • | | | • | • |
| AUClast | Area under the plasma<br>concentration-time curve<br>from time zero to time of last<br>measurable concentration | The area under the concentration-time curve from zero time (pre-dose) to the time of last quantifiable concentration will be calculated using the (specified) trapezoidal method. | h*ng/mL | Y | AUClast | AUCLST | AUC <sub>last</sub> |
| AUC <sub>last</sub> /Dose | Dose-normalised AUC from time zero to last measurable concentration | The dose-normalised AUC from time zero to last measurable concentration will be calculated as AUC <sub>last</sub> /Dose Administered | (h*ng/mL)/mg | Y | - | AUCLSTD | AUC <sub>last</sub> /D |
| $\mathrm{AUC}_{\infty}$ | Area under the plasma concentration-time curve from time zero to infinity | Calculated using the (specified) trapezoidal method for the interval 0 to t <sub>last</sub> (time t <sub>last</sub> is the time at which the last non-zero level was recorded), plus the area under the exponential curve from t <sub>last</sub> to infinity, calculated as follows: | h*ng/mL | Y | AUCINF_pred | AUCIFP | AUC <sub>inf</sub> |

HMR 17 November 2021 Page 47 of 49

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| | | $AUC = \frac{C_t}{\lambda_z} \text{where } c_t \text{ is the}$ predicted value of the concentration at t <sub>last</sub> . | | | | | |
| AUC∞/Dose | Dose-normalised AUC to infinity | Calculated as AUC <sub>∞</sub> /Dose administered | (h*ng/mL)/mg | Y | AUCINF_D_pred | AUCIFPD | AUC <sub>inf</sub> /D |
| %AUCextrap | $\begin{array}{c} \text{Percentage of AUC}_{\infty} \\ \text{extrapolated from from } t_{last} \\ \text{to infinity} \end{array}$ | $\%AUC_{extrap} = \frac{100 \times AUC_{t-\infty}}{AUC_{\infty}}$ | % | N | AUC_%EXTRAP_pred | AUCPEP | %AUCextrap |

HMR 17 November 2021 Page 48 of 49

# Appendix B: Sample page layout

| Population: [Pop] | Page x of y* |
|----------------------------------------------------|---------------|
| Table [number] [title] | |
| Column headers | |
| Main body of output | |
| Source: Listing [16.2.xx] | |
| Footnotes about the table or listing text go here. | |
| Program: [Prog Name] [Date] | HMR 21-001 |
| Produced By: [Username] | IIVIIX 21-001 |

\*y = last page of individual output Font size will be Arial 9.5pt. The following margins will be used: Left: 1", Right: 1", Top: 1", Bottom: 1"



# ASN51-102 (HMR 21-001) SAP v1 (17Nov2021)

Final Audit Report 2021-11-24

Created: 2021-11-18

By: Status: Signed

Transaction ID: CBJCHBCAABAAdXvkO\_3E8PfoQULrGjJ-KjMBj5CZarF6

# "ASN51-102 (HMR 21-001) SAP v1 (17Nov2021)" History

| | 131131-102 (1111111 21-001) 3A1 VI (1 | 11100202 |
|---|---|---|
| 1 | Document created by 2021-11-18 - 8:12:13 AM GMT | |
| <b></b> | Document emailed to 2021-11-18 - 8:13:10 AM GMT | for signature |
| 1 | Email viewed by 2021-11-22 - 8:03:22 AM GMT- IP address: | |
| Ø <sub>B</sub> | Document e-signed by Signature Date: 2021-11-22 - 8:03:47 AM GMT - Time Source: server- IP address | es: |
| <b></b> | Document emailed to | for signature |

Document e-signed by

E-signature obtained using URL retrieved through the Adobe Sign API

Signature Date: 2021-11-24 - 1:55:14 PM GMT - Time Source: server

Agreement completed.

2021-11-24 - 1:55:14 PM GMT